CLINICAL TRIAL: NCT05134857
Title: Zonisamide for the Treatment of Alcohol Use Disorder in the Addiction Neuroclinical Assessment Framework
Brief Title: The Zonisamide and Reinforcement for Reducing Alcohol Use (ZARRA) Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Sterling McPherson, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18520-001
Record Dates: First submitted 2021-10-14; First posted 2021-11-26 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol Use Disorder; Zonisamide; Contingency Management; Incentives for Sobriety
MeSH Terms: conditions — Alcoholism | interventions — Zonisamide

STUDY DESIGN:
Intervention Model Description: A phase II randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZON+ST (Experimental): Zonisamide (ZON) plus standard treatment (ST)
  Interventions: Drug: Zonisamide
- PLO+ST (Placebo Comparator): Placebo (PLO) plus standard treatment (ST)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide — The ZON will be supplied in 100 mg capsules and deposited directly into the TAD device by research staff every 2 weeks. All participants will be told to take 100 mg/day for the first three weeks (Week 1-2 single-blind, placebo-only, induction; end of Week 2, active treatment begins) and increasing by 100 mg/day every other week (Week 4: 200 mg/day; Week 6: 300 mg/day; Week 8: 400 mg/day) up to the target dose of 500 mg/day by Week 10. The participants will be maintained on this dose through Week 14 of active treatment and then tapered off ZON (2 weeks). This dosing schedule is consistent with best practices for ZON. All TAD devices will only dispense the prescribed medication between 4pm and 11pm each night. Participants will be instructed to take the medication at or near bedtime.
  Arms: ZON+ST
Drug: Placebo — The PLO will be supplied at the same schedule and in the same manner (TAD device) as the ZON.
  Arms: PLO+ST

SUMMARY:
A phase II randomized, double-blind, placebo-controlled clinical trial (RCT) to evaluate the ability of zonisamide (ZON) to decrease alcohol use among treatment-seeking adults with an alcohol use disorder (AUD).

DETAILED DESCRIPTION:
This project focuses on the efficacy of a promising pharmacotherapy (ZON) for AUDs using a placebo-controlled design that will rigorously measure alcohol use and medication adherence. Results will guide novel mechanistic targets to better capture the heterogeneity within AUDs. This project will evaluate the ability of ZON to treat the alcohol use disorder.

The investigators hypothesize that the group assigned to ZON associated with the standard treatment (ZON+ST) will yield lower rates of biochemically verified alcohol use, fewer self-reported drinks per day, and fewer heavy drinking days during the 12-week treatment and 1-year follow-up periods, relative to the placebo associated with the standard treatment (PLO+ST) group.

ELIGIBILITY:
Inclusion Criteria:

1. Four or more standard drinks on four or more occasions in the prior 30 days.
2. Seeking AUD treatment.
3. Aged 18-65 years.
4. DSM-5 diagnosis of AUD.
5. Ability to read and speak English.
6. Ability to provide written informed consent.
7. Breath alcohol of 0.00 during informed consent.
8. Provision of at least 1 EtG-positive urine test at any time during the induction period.
9. Non-lactating women of childbearing age using reliable form of birth control with a negative urine pregnancy test at baseline, and
10. Attended at least 4 of 6 visits during the induction period.

Exclusion Criteria:

1. Significant risk of dangerous alcohol withdrawal, defined as a history of alcohol detoxification or seizure in the last 12 months and expression of concern by the participant about dangerous withdrawal;
2. Currently receiving any pharmacotherapy for alcohol or in the past 30 days.
3. Current DSM-5 diagnosis of severe substance use disorder other than nicotine.
4. Suicide attempt in the last 20 years.
5. History of hypersensitivity to sulfonamide medication, Stevens-Johnson Syndrome, penicillin allergy or allergic reaction to any drug
6. Systemic autoimmune disease.
7. History of current seizure disorder (e.g., are they receiving medication currently for their seizures, have they ever been told by their provider that they have epilepsy, or do they have a history of recurring seizures in the last 5 years?).
8. Current clinically significant blood dyscrasia.
9. History of clinically significant renal calculi or renal failure; renal compromise (defined by an elevation of serum creatinine above our laboratory's limit of normal).
10. History of traumatic brain injury (TBI; e.g., ever been told by a provider that they had a moderate or severe TBI, lost consciousness for 30 minutes or longer or had a post-traumatic amnesia lasting a day or longer).
11. Any other current, clinically significant physical disease [i.e., neurologic, renal, rheumatologic, gastrointestinal, hematologic, pulmonary, endocrine, cardiovascular, hepatic, or autoimmune disease] on the basis of medical history, physical examination, or routine laboratory evaluation that, in the context of the study would represent a risk to the subject, or significant laboratory abnormalities related to hepatic function such as marked elevations of hepatic aminotransferase levels (i.e., AST and ALT) or direct bilirubin, and
12. Any other medical or psychiatric condition that Dr. Rodin determines would compromise safe participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Self Reported Alcohol Consumption | 12-week treatment and 1-year follow-up period
  Consumption of alcohol between participants randomized to ZON+ST vs PLO+ST assessed by participant self report (collected 1x weekly from weeks 1-14 and once at weeks 18, 38, and 54).

SECONDARY OUTCOMES:
Change in Biochemically Verified Alcohol Consumption | 12-week treatment and 1-year follow-up period
  Consumption of alcohol between participants randomized to ZON+ST vs PLO+ST assessed by alcohol breathalyzer and biochemical EtG values (collected 3x weekly from weeks 1-6, 1x weekly at weeks 7-14, and once at weeks 18, 38, and 54).

OTHER OUTCOMES:
Adverse Events | 12-week treatment and 1-year follow-up period
  Occurrence of adverse events assessed by SAFETEE (collected 3x weekly at weeks 1-6, 1x weekly at weeks 7-14, and once at weeks 18, 38, and 54).

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is to be shared with NIAAA under their required data archiving procedures.
Supporting Information: CSR
Time Frame: 5-6 years
Access Criteria: Determined by NIAAA data archive policy
URL: https://www.niaaa.nih.gov/research/niaaa-data-archive